CLINICAL TRIAL: NCT05378230
Title: Effects of the Probiotic AB-LIFE on the Amount and Profile of Bile Acids, and the Lipid and Metabolic Profile in Healthy Overweight Subjects.
Brief Title: Probiotic Intervention, Bile Acids and Lipid Metabolism Metabolic Profile in Healthy Overweight Subjects.
Acronym: PROBILIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: AB Biotics, SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IIBSP-PRO-2019-122
Record Dates: First submitted 2022-05-05; First posted 2022-05-18 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Probiotic Intervention
Keywords: Microbiota; Bile acids; Lipids; Inflammation; Metabolism
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: The intervention trial consisted of a single-center, one-arm study with a total duration of 8 weeks, which includes 2-weeks run-in period, 4 week intervention period and 2-weeks post-intervention or wash-out period. The intervention period was divided in 4 periods of 7 days each and the treatment consisted of increasing dose of Lactobacillus plantarum AB-B (CECT 7527, CECT 7528, CECT 7529).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Probiotic mixture (Experimental): Arm that received Lactobacillus plantarum mixture (CECT 7527, CECT 7528 and CECT 7529)
  Interventions: Dietary Supplement: Probiotic preparation of three Lactobacillus plantarum strains (CECT 7527, CECT 7528, CECT 7529)

INTERVENTIONS:
Dietary Supplement: Probiotic preparation of three Lactobacillus plantarum strains (CECT 7527, CECT 7528, CECT 7529) — All subjects were submitted to 4 weeks intervention consisting on a dose-dependent regime of Lactobacillus plantarum AB-B (strains CECT 7527, CECT 7528, CECT 7529; AB-LIFE). Before starting the intervention period, all subjects were submitted to a 2-weeks run-in period. During the wash-in and intervention-periods, participants were instructed to maintain their habitual dietary habits and to continue their normal pattern of physical activity throughout the study period.
  Treatments during the intervention period were: Week 1: 1 capsule/day taken during breakfast; Week 2: 2 capsules / day at- breakfast; Week 3: 2 capsules at breakfast and 1 at dinner; Week 4: 2capsules at breakfast and 2 capsules at dinner. Each capsule contains 1.2x10^9 cfu (colony forming units) in a 1: 1: 1 ratio of the three strains.
  Other Names: AB-LIFE

SUMMARY:
Moderate hypercholesterolemia, metabolic alterations derived from overweight or obesity, and consequently and their related cardiovascular risks can be reduced through changes in lifestyle. A growing body of evidence shows a relationship between hypercholesterolemia and dysfunction of the gut microbiota.

Gut microbiota is considered a keystone in maintaining the health condition of the host through multiple mechanisms affecting different metabolic processes, including lipid metabolism and cholesterol-related pathways. Bile acids (BA) are cholesterol-derived compounds synthesized in the liver and metabolized upon modification by gut bacteria once they reach the colon.

Conversely, BAs shape the composition and function of the intestinal microbiota. This mutual interplay between BAs and gut microbiota regulates many physiological processes, including the lipid, carbohydrate and energy metabolism of the host.

Previous studies based on Lactobacillus plantarum have shown 3 strains CECT 7527, 7528, and 7529 with the ability to adhere to the intestinal mucosa with very low toxicity, what makes them susceptible to be used as a probiotic. The lipid-lowering effect of the 3 bacteria strains was already evidenced in previous preclinical studies in animal models and clinical studies in hypercholesterolemic subjects. Up to now, however, little is known about the effects of the 3- combined Lactobacillus plantarum strains on levels and profile of bile acids in healthy overweight subjects, otherwise at low cardiovascular risk.

The aim of this study is to explore on the mechanism of action of a Lactobacillus plantarum mixture (CECT 7527, CECT 7528 and CECT 7529) and evaluate the effect of this probiotic formulation on BA profile as well as on plasma lipids and other related biomarkers when administered in a dose-dependent regime in a cohort of overweight subjects.

The probiotic product was administrated for 4 weeks with a weekly dose-regime of 2x, 3x, and 4x, respectively, in the second, third, and fourth week in relation to the first week. The effects were evaluated on: (1) level and profile of bile acids in plasma and feces, (2) plasma lipid/lipoprotein and fatty acid profile and (3) endocrine hormones, glucose metabolism and inflammatory markers in plasma.

DETAILED DESCRIPTION:
Sample size (N=20) was calculated according results of previous studies on plasma bile acids. The study refers to healthy overweight [body mass index (BMI) 25.0-29.9 kg/m2] adult men (N=10) and women (N=10) between the ages of 25 and 60 years.

The study was approved by the Human Ethical Review Committee of the Hospital Sant Pau in Barcelona (register number: 20/029). Informed written consent was obtained from all participants before their inclusion in the study. To confirm health status, all subjects underwent a complete physical examination conducted by the study physician.

The study lasted 6 weeks that were structured in:

* 2 weeks of run-in.
* 4 weeks of intervention period divided into 4 phases of 7 days. During the intervention period, Lactobacillus plantarum capsules were consumed according to the following pattern:

  * Days 0-6: 1 capsule/day
  * Days 7-13: 2 capsules/day
  * Days 14-20: 3 capsules/day
  * Days 21-27: 4 capsules/day

The volunteers visited the center at the beginning of each phase of the intervention period (Days 0, 7, 14 and 21) and at the end of the intervention period (Day 28).

Dietary habits were collected. Compliance was monitored by weekly telephone contact with participants and interviewing them at the end of each intervention period. Blood samples were collected early at the morning after twelve-hour fasting at baseline and at the end of each intervention phase. Blood samples were used for determining all variables of the study. Stool samples were obtained at baseline and after 28 days intervention for the study of bile acids, fatty acids and microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass index (BMI): Between 25 and 30 Kg / m2

Exclusion Criteria:

* Eating disorders.
* Subjects with cardiovascular risk factors such as hypercholesterolemia (genetic or secondary), hypertension and diabetes, treated pharmacologically.
* History of ischemic heart disease (and / or previous angina or AMI) or arrhythmia (current or previous).
* Previous strokes and / or peripheral vascular disease.
* Alcohol consumption greater than 60 gr / day.
* Kidney failure (creatinine> 2 mg / dl).
* Presence of neoplasia.
* Presence of systemic disease.
* Psychiatric illness under treatment with psychotropics.
* Unstabilized thyroid disease.
* Having followed or being following a hypocaloric diet or regularly consumed dietary supplements for weight or constipation or cholesterol control (plant sterols, soy lecithin, omega-3 fatty acids) for 2 months prior to inclusion in the study.
* Pregnancy or breastfeeding.
* In current treatment with non-steroidal anti-inflammatory drugs, antiplatelet agents, fibrates or statins.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-11-28 (Actual); Study Completion 2022-02-21 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Lipid profile at 7 days | At days 0 and 7
  By standardized biochemical techniques
Change from Baseline Lipid profile at 14 days | At days 0 and 14
  By standardized biochemical techniques
Change from Baseline Lipid profile at 21 days | At days 0 and 21
  By standardized biochemical techniques
Change from Baseline Lipid profile at 28 days | At days 0 and 28
  By standardized biochemical techniques
Change from Baseline Serum bile acids at 14 days | At days 0 and 14
  By ultra-high performance liquid chromatography - mass spectrometry (UHPLC-MS)
Change from Baseline Serum bile acids at 28 days | At days 0 and 28
  By ultra-high performance liquid chromatography - mass spectrometry (UHPLC-MS)
Change from Faecal bile acids at 28 days | At days 0 and 28
  By ultra-high performance liquid chromatography - mass spectrometry (UHPLC-MS)
Change from Baseline Serum fatty acids at 14 days | At days 0 and 14
  By ultra-high performance liquid chromatography - mass spectrometry (UHPLC-MS)
Change from Baseline Serum fatty acids at 28 days | At days 0 and 28
  By ultra-high performance liquid chromatography - mass spectrometry (UHPLC-MS)
Change from Baseline Faecal fatty acids at 28 days | At days 0 and 28
  By ultra-high performance liquid chromatography - mass spectrometry (UHPLC-MS)
Change from Baseline Serum lipoprotein profile at 14 days | At days 0 and 14
  By nuclear magnetic resonance (NMR)
Change from Baseline Serum lipoprotein profile at 28 days | At days 0 and 28
  By nuclear magnetic resonance (NMR)
Change from Baseline Plasmatic endocrine hormones and metabolic markers at 14 days | At days 0 and 14
  By Enzyme-Linked immunosorbent Assay (ELISAs)
Change from Baseline Plasmatic endocrine hormones and metabolic markers at 28 days | At days 0 and 28
  By Enzyme-Linked immunosorbent Assay (ELISAs)

SECONDARY OUTCOMES:
Change from Baseline Plasmatic Inflammatory markers at 14 days | At days 0 and 14
  By standardized biochemical techniques and Multiplex for Luminex Immunoassays
Change from Baseline Plasmatic Inflammatory markers at 28 days | At days 0 and 28
  By standardized biochemical techniques and Multiplex for Luminex Immunoassays
Change from Baseline LDL susceptibility to oxidation and HDL antioxidant capacity at 14 days | At days 0 and 14
  By conjugated dienes measurement and by Total radical-trapping antioxidant potential (TRAP) respectively
Change from Baseline LDL susceptibility to oxidation and HDL antioxidant capacity at 28 days | At days 0 and 28
  By conjugated dienes measurement and by Total radical-trapping antioxidant potential (TRAP) respectively
Change from Baseline Serum Vitamin D and thyroid hormones (TSH, T3 & T4) at 14 days | At days 0 and 14
  By Liquid Chromatography with tandem mass spectrometry (LC-MS/MS) and by chemoluminescence immunoassays respectively
Change from Baseline Serum Vitamin D and thyroid hormones (TSH, T3 & T4) at 28 days | At days 0 and 28
  By Liquid Chromatography with tandem mass spectrometry (LC-MS/MS) and by chemoluminescence immunoassays respectively

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Recerca-Hospital Santa Creu I Sant Pau, Barcelona, Spain

REFERENCES:
- [Derived] Padro T, Santisteban V, Huedo P, Puntes M, Aguilo M, Espadaler-Mazo J, Badimon L. Lactiplantibacillus plantarum strains KABP011, KABP012, and KABP013 modulate bile acids and cholesterol metabolism in humans. Cardiovasc Res. 2024 May 29;120(7):708-722. doi: 10.1093/cvr/cvae061. PMID 38525555